CLINICAL TRIAL: NCT07100054
Title: Pharmacogenomic and Circulating Biomarkers for Predicting Toxicity or Suboptimal Benefit From Small Molecule Kinase Inhibitor Therapy
Brief Title: Pharmacogenomic and Circulating Biomarkers for CDK4/6 Inhibitors
Status: Enrolling by invitation | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Kim, Clinical Pharmacologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: P.CTP.1262
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: CDK4/6 Inhibitor; Breast Cancer; CYP3A4 Protein, Human; Drug Interaction; Pharmacogenetic Testing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected at each in-person appointment for extraction of DNA (genotype) and plasma (drug level and biomarker analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Whole gene sequencing — Whole gene sequencing of CYP3A4 and PXR
Other: Drug-drug interaction analysis — Evaluating potential drug interactions with CYP3A4 inhibitors and inducers
Other: Biomarker analysis — Determination of circulating CYP3A4 mRNA, and 4b-hydroxycholesterol

SUMMARY:
The goal of this research study is to reduce adverse effects of anti-cancer medications known as kinase inhibitors, while preserving their therapeutic benefits.

There have been major advances in the way cancers are treated. A class of drugs known as kinase inhibitors have proven to be highly effective for the treatment of cancers, including lung, kidney, gastrointestinal, and breast cancers. However, kinase inhibitor medications are well known for having unpredictable side effects.

The body breaks down (metabolizes) medications such as kinase inhibitors using an enzyme known as cytochrome P450 3A4 (CYP3A4). CYP3A4 is the most important drug metabolizing enzyme in humans due to the fact that it is involved in the metabolism of nearly half of all prescribed medications and almost all of the currently prescribed kinase inhibitors. Among patients, there can be nearly 400 times difference in how efficiently CYP3A4 metabolizes drugs. Remarkably, very little is known about the role of genetic differences in CYP3A4 and a gene known as pregnane X receptor (PXR). PXR serves as a sensor for drugs in the body and helps to regulate how much CYP3A4 is made. Currently, there are no predictive biomarkers, whether in genes (genomic) or circulating in blood (endogenous) that could aid treating oncologists with regards predicting adverse effects or suboptimal response to this important class of anticancer drugs.

The goal is to carry out DNA sequencing for genetic changes in CYP3A4 and PXR to assess differences in enzyme activity of not only common, but also rare genetic variants. CYP3A4 activity will be determined in participants blood samples based on break down products of the drug tamoxifen as well as cholesterol, the latter called 4β-hydroxycholesterol, both known to be influenced by the CYP3A4 enzyme. Since cholesterol is naturally made in the body, comparing blood cholesterol to 4β-hydroxycholesterol levels will be a biomarker of CYP3A4 metabolic activity that can be measured in anyone. Furthermore, circulating CYP3A4 messenger RNA from human blood will be measured as another independent marker of CYP3A4 gene expression. A model will be generated that includes these biomarkers of CYP3A4 expression and function, as well as genetic variation in CYP3A4 and PXR, that will aid in better identifying which patients may be at risk for loss of benefit or toxicity from kinase inhibitor therapy. This model will be evaluated in 100 breast cancer patients undergoing chemotherapy with kinase inhibitors, namely cyclin-dependent kinases CDK4 and CDK6 inhibitor (abemaciclib, ribociclib or palbociclib), as such kinase inhibitors are widely prescribed for breast cancer and are known to be broken down by CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* female
* breast cancer diagnosis
* over 18 years of age
* indication for a CDK4/6 inhibitor treatment
* proficient in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational cohort will consist of female adult cancer patients routinely seen at the London Regional Cancer Program for breast cancer chemotherapy. Patients must be starting or currently on the CDK4/6 inhibitors abemaciclib, ribociclib and palbociclib for the treatment of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Predictive model for CDK4/6 inhibitor concentrations | From enrollment to 3 months
  A linear mixed effect model will be applied using CDK4/6 inhibitor levels considering the following independent variables: sex, age, body surface area, height, weight, serum creatinine, drug dose, CYP3A4 and PXR genotype (any impaired-function SNV carrier vs. normal function SNV carrier status/wildtype as per in vitro analysis), CYP3A4 mRNA and 4β-hydroxycholesterol. The model that best describes the fit of CDK4/6 pharmacokinetics will be selected.

SECONDARY OUTCOMES:
Patient reported outcomes | From enrollment to 3 months
  Evaluate the association in patient reported outcomes in the EORTC QLG Core Questionnaire (EORTC QLC-C30) with drug concentrations and/or treatment-related toxicity using common terminology criteria for adverse events (CTCAE). CTCAE is graded on a scale from 1 to 5 with a higher number indicating more toxicity. The EORTC QLC-C30 is a 30-item instrument to assess quality of life. The first 28 items are rated on a scale from 1 to 4 with a higher score indicating worse outcome. The last 2 items are rated on a scale of 1 to 7 with a higher number indicating better health and quality of life.
Patient reported outcomes | From enrollment to 3 months
  Evaluate the association in patient reported outcomes using the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-BR42) with drug concentrations and/or treatment-related toxicity using common terminology criteria for adverse events (CTCAE). The CTCAE is graded on a scale from 1 to 5 with a higher number indicating more toxicity. The QLQ-BR42 is a 42 item scale rated from 1 to 4 with a higher number indicating a worse outcome.

OTHER OUTCOMES:
Exploratory breast cancer outcomes | From enrollment to 3 months
  Evaluate efficacy of CDK4/6 by examining breast cancer outcomes, including invasive disease-free survival (IDFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No